CLINICAL TRIAL: NCT01494402
Title: A Phase I, Open Label, Randomized, Single Center, 2 Way Crossover Bioequivalence Study Comparing D961S (a Fixed-dose Combination Capsule of Esomeprazole 20 mg and Acetylsalicylic Acid 81 mg) With a Free Combination of Esomeprazole Capsule 20 mg + Buffered Acetylsalicylic Acid Tablet 81 mg After Repeated Oral Administration in Japanese Healthy Male Subjects
Brief Title: Study to Assess the Bioequivalence Between D961S and Esomeprazole/Buffered Acetylsalicylic Acid (ASA) in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D961SC00001
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Bioequivalence Study
Keywords: Healthy volunteer, Japanese males, homo-EM
MeSH Terms: interventions — Esomeprazole

ARMS (2):
- D961S (Experimental): 2 way crossover
  Interventions: Drug: D961S
- esomeprazole + buffered acetylsalicylic acid (Experimental): 2 way crossover
  Interventions: Drug: Esomeprazole; Drug: Buffered acetylsalicylic acid

INTERVENTIONS:
Drug: D961S — Oral gelatine capsule
  Arms: D961S
Drug: Esomeprazole — Oral HPMC capsule
  Other Names: Nexium® capsule 20 mg
  Arms: esomeprazole + buffered acetylsalicylic acid
Drug: Buffered acetylsalicylic acid — Tablet
  Other Names: Bufferin Combination Tablet A81
  Arms: esomeprazole + buffered acetylsalicylic acid

SUMMARY:
The purpose of this study is to assess bioequivalence between D961S and esomeprazole/buffered ASA, safety, tolerability of esomeprazole in combination with ASA and pharmacokinetics (PK) of D961S, esomeprazole and buffered ASA following repeated administration in healthy male Japanese subjects.

DETAILED DESCRIPTION:
A Phase I, Open label, Randomized, Single center, 2 way Crossover Bioequivalence Study Comparing D961S (a Fixed-dose Combination Capsule of Esomeprazole 20 mg and Acetylsalicylic Acid 81 mg) with a Free Combination of Esomeprazole Capsule 20 mg + Buffered Acetylsalicylic Acid Tablet 81 mg After Repeated Oral Administration in Japanese Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males 20-45 years of age
* Classified as homo-EM
* Negative for HIV, Hepatitis B, Hepatitis C and syphilis
* Body Mass Index (BMI=weight/height2) 19-27 (kg/m2)
* Body weight 50-85 kg

Exclusion Criteria:

* Significant clinical illness from 2 weeks preceding the pre-entry visit to the randomization
* Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease
* Need for concomitant medication in the study
* Past or present NSAIDs induced asthma
* History of bleeding diathesis

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Description of bioequivalence of D961S to combination of esomeprazole + buffered ASA in terms of Area under the plasma concentration(AUCτ). | Baseline, which is 30 minutes before dose at day 5 of treatment period, till day 6
  All PK variables at each time point will be listed by subject and summarised for each treatment using appropriate descriptive statistics.
Description of bioequivalence of D961S to combination of esomeprazole + buffered ASA in term maximum plasma concentration (Cmax,ss) | Baseline, which is 30 minutes before dose at day 5 of treatment period, till day 6
  All PK variables at each time point will be listed by subject and summarised for each treatment using appropriate descriptive statistics.

SECONDARY OUTCOMES:
Description of D961S PK profile comparing to esomeprazole and ASA combination in terms of AUC0-t,ss, mean residence time (MRT), time to reach Cmax (tmax,ss) and t1/2,ss of esomeprazole and ASA, and AUCτ, Cmax,ss, AUC0-t,ss, MRT, tmax,ss and t1/2,ss of SA | Baseline, which is 30 minutes before dose at day 5 of treatment period, till day 6
  All PK variables and plasma concentrations of esomeprazole, ASA and SA at each time point will be listed by subject and summarised for each treatment using appropriate descriptive statistics.
Description of Safety and tolerability profile of esomeprazole in combination with ASA in terms of adverse events, clinical laboratory tests, blood pressure, pulse rate and body temperature. | Pre-entry, Day 5 of treatment period and follow up (5-7 days after last dose)
  Descriptive statistics will be provided for all safety variables, and the analyses will be performed according to the actual treatment. No formal comparison will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Study site, Hakata, Fukuoka, Japan